CLINICAL TRIAL: NCT01375049
Title: Open-Label Phase 2 Trial to Evaluate the Safety and Efficacy of Aztreonam 75 mg Powder and Solvent for Nebuliser Solution/Aztreonam for Inhalation Solution (AZLI) in Pediatric Patients With Cystic Fibrosis (CF) and New Onset Lower Respiratory Tract Culture Positive for Pseudomonas Aeruginosa (PA)
Brief Title: Aztreonam Lysine for Pseudomonas Infection Eradication Study
Acronym: ALPINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-205-0162
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; CF; PA; Pseudomonas aeruginosa; AZLI; aztreonam
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Aztreonam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aztreonam for Inhalation Solution (AZLI) (Experimental): Participants will receive one 28-day course of AZLI, then will be followed for a 24-week period (through Day 196).
  Interventions: Drug: Aztreonam for Inhalation Solution (AZLI)

INTERVENTIONS:
Drug: Aztreonam for Inhalation Solution (AZLI) — AZLI 75 mg administered 3 times daily via the investigational eFlow® nebulizer
  Other Names: Cayston®

SUMMARY:
This is an open-label, multi-center study in pediatric patients age 3 months to less than 18 years with cystic fibrosis (CF) and newly detected Pseudomonas aeruginosa (PA) pulmonary colonization/infection. All eligible participants will be treated with a 28-day course of Aztreonam for Inhalation Solution (AZLI) 75 mg 3 times daily. After completion of study drug, subjects will be followed up through Day 196 for safety and recurrence of PA.

The primary objective is to evaluate the proportion of participants with PA-negative cultures at all time points during a 6-month monitoring period (through Day 196) after cessation of AZLI treatment. Microbiological cultures will be obtained at Baseline, Day 28 (end of AZLI treatment), Day 56 (1 month after completing AZLI treatment), Day 112 (3 months after completing AZLI treatment), and Day 196 (6 months after completing AZLI treatment).

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 3 months to less than 18 years
* Diagnosis of CF as determined by the 1997 CF Consensus Conference criteria:
* Documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test OR
* Abnormal nasal transepithelial potential difference test OR
* Two well-characterized, disease-causing genetic mutations in the CF transmembrane conductance regulator (CFTR) gene AND
* One or more clinical features consistent with CF
* Documented new onset of positive lower respiratory tract culture (e.g., throat swab, sputum, or BAL) for PA within 30 days of study entry (prior to screening visit) defined as either first lifetime documented PA-positive culture OR PA recovered after at least a 2 year history of PA-negative respiratory cultures (at least 2 cultures per year)
* Forced expiratory volume in 1 second (FEV1) ≥ 80% predicted at screening visit (subjects ≥ 6 years of age)
* Clinically stable with no evidence of significant respiratory symptoms or, if obtained for clinical evaluation, no chest radiograph findings at screening that would have required administration of IV antipseudomonal antibiotics, oxygen supplementation, or hospitalization.
* All sexually active females who were of childbearing potential must agree to use a highly effective method of contraception during heterosexual intercourse throughout the study. Females utilizing hormonal contraceptives as a birth control method must have used the same method for at least 3 months prior to study drug dosing.
* Males must agree to use barrier contraception (condom with spermicide) during heterosexual intercourse from screening through to study completion and for 90 days from the last dose of study investigational medicinal product
* Participants and/or parent/guardian must be able to give written informed consent prior to any study related procedure

Exclusion Criteria:

* Use of IV or inhaled antipseudomonal antibiotics within 2 years of study entry (screening visit)
* Use of oral antipseudomonal antibiotics within 30 days of study entry (screening visit)
* History of sputum or throat swab culture yielding Burkholderia spp. within 2 years prior to screening visit
* History of local or systemic hypersensitivity to monobactam antibiotics
* History of intolerance to inhaled short acting beta 2 agonists
* History of lung transplantation
* History of AZLI (or Cayston®) administration
* Administration of any investigational drug or device within 28 days prior to screening visit or within 6 half-lives of the investigational drug (whichever is longer)
* Current use of oral corticosteroids in doses exceeding the equivalent of 10 mg prednisone per day or 20 mg prednisone every other day
* Current requirement for daily continuous oxygen supplementation or requirement of more than 2 L/minute at night
* Hospitalization for pulmonary-related illness within 28 days prior to screening visit
* Changes in or initiation of chronic azithromycin treatment within 28 days prior to screening visit
* Changes in antimicrobial, bronchodilator (BD), corticosteroid, dornase alfa, or hypertonic saline medications within 7 days prior to screening visit; for participants on a stable regimen of hypertonic saline (28 days on/28 days off), beginning or ending a cycle of hypertonic saline is allowed
* Changes in physiotherapy technique or schedule within 7 days prior to screening visit
* Abnormal renal or hepatic function results at most recent test within the previous 12 months, defined as:
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times upper limit of normal (ULN), or
* Serum creatinine > 2 times ULN for age
* Pregnant or lactating females; a negative urine pregnancy test is required for all females of childbearing potential (unless surgically sterile), and confirmatory serum pregnancy test in the event of an initial positive urine test result
* Any serious or active medical or psychiatric illness (including drug or alcohol abuse), which in the opinion of the investigator, would interfere with treatment, assessment, or compliance with the protocol
* Presence of a condition or abnormality that would compromise the patient's safety or the quality of study data, in the opinion of the investigator

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bresnik, MD, Study Director — Gilead Sciences
Locations (58):
- United States (23):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Nemours Children's Clinic- Jacksonville, Jacksonville, Florida
  - Nemours Childrens Clinic Orlando, Orlando, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Cohen Children's Medical Center of NY, Great Neck, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Toledo Children's Hospital CF Research Center, Toledo, Ohio
  - PennState Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Medizinische Universität Innsbruck Abt. für Kinder- und Jugendheilkunde, Pädiatrie III (Zystische Fibrose), Innsbruck, Austria
- Belgium (4):
  - Hôpital Universitaire des Enfants Reine Fabiola Brussels, Brussels
  - Paediatrics, University Hospital Brussels (UZB), Brussels
  - Pediatric Respiratory Department, Ghent University Hospital, Ghent
  - Pediatric Pulmonology, Dept Pediatrics University Hospital Gasthuisberg, Leuven
- France (7):
  - CHU de Boredaux Hôpital des Enfants - Pellegrin CEDRE, Bordeaux
  - CRCM mixte / CHU ESTAING, Clermont-Ferrand
  - CHI de Créteil Departement pediatrie, Créteil
  - Centre hospitalier Robert Bissons CRCM - service pédiatrie, Lisieux
  - Service pédiatrie II Hôpital Necker Enfants Malades, Paris
  - Hopital Robert Debre, Paris
  - Centre de Ressources et de Compétences sur la Mucoviscidose ( CRCM), Roscoff, France, Roscoff
- Germany (7):
  - Charité Campus Virchow Klinikum, Universitätsmedizin Berlin, Klinik für Pädiatrie mit Schwerpunkt Pneumologie/Immunolgie Prof. Wahn, Berlin
  - Klinik fur Kinder- und Jugendmedizinim St Josef-Hopsital, Bochum
  - Universitätsklinikum Essen, Zentrum für Kinderheilkunde - Abteilung Allg. Kinderheilkunde/Neuropaediatrie, Erlangen
  - Universitaetsklinikum Bonn-Zentrum fuer Kinderheikunde, Essen
  - Christiane Herzog CF-Center, Goethe University Hospital, Frankfurt
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - University Children's Hospital, Tübingen
- Italy (5):
  - Azienda Ospedaliero-Universitaria di Catania, Dipartimento di Pediatria, UO Broncopneumologia Pediatrica, Catania
  - Cystic Fibrosis Centre Paediatric Department, A. Meyer Children Hospital Florence, Florence
  - Universita' Federico II di Napoli, Napoli
  - Fondazione IRCCS, Ospedale Pediatrico, Bambino Gesu' di Roma, Rome
  - Centro Fibrosi Cistica di Verona, Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Netherlands (2):
  - Division of Respiratory Medicine and Allergology, Department of Pediatrics, Erasmus MC-Sophia Children's Hospital, Rotterdam, The Netherlands, Rotterdam
  - Longziekten Universitair Medisch (PEDIATRIC), Ultrecht, Utrecht
- Poland (4):
  - ISPL Centrum Medyczne, Bialystok
  - Specjalistyczny Zespół Opieki Zdrowotnej nad Matką i Dzieckiem, Poradnia Leczenia Mukowiscydozy, Gdansk
  - Instytut Gruźlicy i Chorób Płuc, Klinki Pneumologii i Mukowiscydozy, Rabka-Zdrój
  - Instytut Matki i Dziecka Klinika Pediatrii, Warsaw
- Spain (5):
  - Hospital Vall D' Hebron Pediatric Pneunmonology and Cystic Fibrosis Clinic, Barcelona
  - Hospital infantil Universitario Niño Jesus, Servicio de Neumología Pediatrica, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Infantil La Paz, Madrid
  - Hospital Materno-Infantil Carlos Haya, Servicio de Neumología Pediatrica, Málaga

REFERENCES:
- [Derived] Tiddens HA, De Boeck K, Clancy JP, Fayon M, H G M A, Bresnik M, Derchak A, Lewis SA, Oermann CM; ALPINE study investigators. Open label study of inhaled aztreonam for Pseudomonas eradication in children with cystic fibrosis: The ALPINE study. J Cyst Fibros. 2015 Jan;14(1):111-9. doi: 10.1016/j.jcf.2014.06.003. Epub 2014 Aug 1. PMID 25091537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 46 study sites in the United States and Europe. The first participant was screened on 04 October 2011. The last participant observation occurred on 29 May 2013.
Pre-assignment Details: 109 participants were screened; 105 participants were enrolled and treated, and comprise the Safety Analysis Set and the Full Analysis Set.
Groups:
- AZLI: Participants received one 28-day course of Aztreonam for Inhalation Solution (AZLI), then were followed for a 24-week period (through Day 196). AZLI 75 mg was administered 3 times daily via the investigational eFlow® nebulizer.
Period: Overall Study
Arm/Group | AZLI
Started | 105
Completed | 55
Not Completed | 50
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Protocol-Specified Withdrawal Criteria | 45

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug
Groups:
- AZLI: Participants received one 28-day course of AZLI, then were followed for a 24-week period (through Day 196). AZLI 75 mg was administered 3 times daily via the investigational eFlow® nebulizer.
Arm/Group | AZLI
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.26 (4.743)
Age, Customized [Number; unit: participants]
  3 months to < 2 years | 24
  ≥ 2 years to < 6 years | 25
  ≥ 6 years to < 18 years | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 58
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Black or African Heritage | 1
  White | 99
  Other | 2
  Not Permitted to be Recorded | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 5
  Not Hispanic | 93
  Not Permitted to be Recorded | 7
Region of Enrollment [Number; unit: participants]
  France | 12
  United States | 56
  Spain | 6
  Poland | 3
  Belgium | 11
  Austria | 3
  Netherlands | 5
  Germany | 4
  Italy | 5
Weight [Mean (Standard Deviation); unit: kg] | 24.8 (15.69)
Height [Mean (Standard Deviation); unit: cm] | 113.9 (33.02)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 17.1 (2.57)
Presence of Pseudomonas aeruginosa (PA) [Number; unit: participants] — Of the 105 participants in the safety analysis set, 3 participants did not provide baseline samples (ie, oropharyngeal swab sample). All participants had a positive PA culture within 30 days of baseline.
  participants
    Present at baseline | 45
    Absent at baseline | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With PA-negative Cultures at All Time Points After Cessation of Active Treatment (Evaluable Analysis Set)
Description: The percentage of participants with PA-negative cultures at all time points after cessation of active treatment at Day 28 (assessed at Days 56, 112, and 196) was summarized for the Evaluable Analysis Set.
Time Frame: Day 28 to Day 196
Population: Evaluable Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- AZLI - Evaluable Analysis Set: Participants received one 28-day course of AZLI, then were followed for a 24-week period (through Day 196). AZLI 75 mg was administered 3 times daily via the investigational eFlow® nebulizer.
  The Evaluable Analysis Set consists of participants who completed study drug and did not receive an additional antipseudomonal antibiotic during the 28-day AZLI treatment course, and either completed the study through Day 196 with PA-negative cultures at every visit without the use of additional antipseudomonal antibiotics from Day 28 through Day 196 or had evidence of a positive PA-positive culture from Day 28 through Day 196.
Arm/Group | AZLI - Evaluable Analysis Set
Number analyzed (Participants) | 79
percentage of participants | 58.2 [47.4 to 69.1]

2. Secondary Outcome: Change From Baseline in FEV1% Predicted
Description: Spirometry assessments were performed only in participants ≥ 6 years of age. Forced expiratory volume in 1 second (FEV1) % predicted was defined as FEV1 of the participant divided by the average FEV1 in the population for any person of similar age, sex and body composition.
Time Frame: Baseline to Days 28, 56, 112, and 196
Population: Participants in the Sensitivity Analysis Set ≥ 6 years of age with available data for this assessment were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of FEV1% predicted
Groups:
- AZLI - Met Primary Efficacy Endpoint: This group included participants who met the primary efficacy endpoint, defined as having PA-negative cultures at all time points after cessation of active treatment through Day 196.
  Participants received one 28-day course of AZLI, then were followed for a 24-week period (through Day 196). AZLI 75 mg was administered 3 times daily via the investigational eFlow® nebulizer.
- AZLI - Did Not Meet Primary Efficacy Endpoint: This group included participants who did not meet the primary efficacy endpoint, defined as having any PA-positive culture at Day 28 through Day 196 or having used anti-PA antibiotics through Day 196.
  Participants received one 28-day course of AZLI, then were followed for a 24-week period (through Day 196). AZLI 75 mg was administered 3 times daily via the investigational eFlow® nebulizer.
Arm/Group | AZLI - Met Primary Efficacy Endpoint | AZLI - Did Not Meet Primary Efficacy Endpoint
Number analyzed (Participants) | 25 | 27
percentage of FEV1% predicted
  Change at Day 28 (n=25 [met], 26 [did not meet]) | -0.23 (10.373) | -0.38 (12.347)
  Change at Day 56 (n=25 [met], 26 [did not meet]) | -0.20 (10.949) | -4.24 (7.513)
  Change at Day 112 (n=25 [met], 19 [did not meet]) | 0.32 (9.830) | -5.10 (7.948)
  Change at Day 196 (n=25 [met], 8 [did not meet]) | -2.47 (8.895) | -8.85 (11.510)

3. Secondary Outcome: Change From Baseline in CFQ-R RSS Score
Description: Respiratory symptoms (eg, coughing, congestion, wheezing) were assessed with the Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Symptoms Scale (RSS) only in participants ≥ 6 years of age. The range of scores (units) is 0 to 100 with higher scores indicating fewer symptoms.
Time Frame: Baseline to Days 28, 56, 112, and 196
Population: Participants in the Sensitivity Analysis Set ≥ 6 years of age with available data for this assessment were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AZLI - Met Primary Efficacy Endpoint | AZLI - Did Not Meet Primary Efficacy Endpoint
Number analyzed (Participants) | 25 | 31
units on a scale
  Change at Day 28 (n=24 [met], 29 [did not meet]) | 8.33 (15.883) | 5.36 (8.937)
  Change at Day 56 (n=24 [met], 27 [did not meet]) | 6.37 (16.433) | 6.17 (11.040)
  Change at Day 112 (n=24 [met], 21 [did not meet]) | 5.79 (14.397) | 1.46 (14.636)
  Change at Day 196 (n=24 [met], 10 [did not meet]) | 6.13 (18.002) | 5.83 (9.663)

4. Secondary Outcome: Percentage of Participants With PA-negative Cultures
Description: The percentage of participants with a PA-negative culture was summarized at each visit.
Time Frame: Days 28, 56, 112, and 196
Population: Participants from the Full Analysis Set who completed study drug and did not receive an additional antipseudomonal antibiotic during the 28-day AZLI treatment course were included in the analysis at all time points.
Measure: Number; unit: percentage of participants
Arm/Group | AZLI
Number analyzed (Participants) | 101
percentage of participants
  Day 28 | 89.1
  Day 56 | 75.2
  Day 112 | 63.4
  Day 196 | 47.5

5. Secondary Outcome: Use of Additional (Non-study) Antipseudomonal Antibiotics
Description: The percentage of participants who used additional (non-study) antipseudomonal antibiotics (an indication of PA exacerbation) while on treatment and posttreatment was summarized.
Time Frame: Baseline to Day 196
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | AZLI
Number analyzed (Participants) | 105
percentage of participants
  On-treatment | 1.9
  Posttreatment | 43.8

6. Secondary Outcome: Change From Baseline in Weight
Time Frame: Baseline to Days 28, 56, 112, and 196
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | AZLI
Number analyzed (Participants) | 105
kg
  Change at Day 28 (On-Treatment, n = 104) | 0.3 (0.70)
  Change at Day 56 (Posttreatment, n = 101) | 0.5 (0.72)
  Change at Day 112 (Posttreatment, n = 90) | 0.8 (1.02)
  Change at Day 196 (Posttreatment, n = 69) | 1.5 (3.8)

7. Secondary Outcome: Change From Baseline in Height
Time Frame: Baseline to Days 28, 56, 112, and 196
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AZLI
Number analyzed (Participants) | 105
cm
  Change at Day 28 (On-Treatment, n = 104) | 0.6 (0.87)
  Change at Day 56 (Posttreatment, n = 101) | 1.4 (1.27)
  Change at Day 112 (Posttreatment, n = 90) | 2.6 (2.00)
  Change at Day 196 (Posttreatment, n = 69) | 4.5 (2.86)

8. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Time Frame: Baseline to Days 28, 56, 112, and 196
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | AZLI
Number analyzed (Participants) | 105
kg/m^2
  Change at Day 28 (On-Treatment, n = 104) | 0.1 (0.57)
  Change at Day 56 (Posttreatment, n = 101) | 0.1 (0.71)
  Change at Day 112 (Posttreatment, n = 90) | 0.0 (0.97)
  Change at Day 196 (Posttreatment, n = 69) | 0.0 (0.93)

9. Secondary Outcome: Pharmacokinetics (PK) Peak and Trough Plasma Concentrations of Aztreonam
Description: The plasma concentration of aztreonam for participants < 6 years of age was obtained 1 hour after the first dose of AZLI on Day 1 and immediately prior to the last dose of AZLI on Day 28.
Time Frame: Day 1 (1 hour postdose) and Day 28 (immediately prior to dosing)
Population: Participants in the Full Analysis Set < 6 years of age with evaluable PK profiles were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AZLI
Number analyzed (Participants) | 49
ng/mL
  Day 1 (1 hour postdose, n = 40) | 578 (560.0)
  Day 28 (immediately prior to dosing, n = 43) | 125 (166.3)

10. Primary Outcome: Percentage of Participants With PA-negative Cultures at All Time Points After Cessation of Active Treatment (Sensitivity Analysis Set)
Description: The percentage of participants with PA-negative cultures at all time points after cessation of active treatment at Day 28 (assessed at Days 56, 112, and 196) was summarized for the Sensitivity Analysis Set.
Time Frame: Day 28 to Day 196
Population: Sensitivity Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- AZLI - Sensitivity Analysis Set: Participants received one 28-day course of AZLI, then were followed for a 24-week period (through Day 196). AZLI 75 mg was administered 3 times daily via the investigational eFlow® nebulizer.
  The Sensitivity Analysis Set consists of participants who completed study drug and did not receive an additional antipseudomonal antibiotic during the 28-day AZLI treatment course, and either completed the study through Day 196 with PA-negative cultures at every visit without the use of additional antipseudomonal antibiotics from Day 28 through Day 196 or had evidence of a PA-positive culture from Day 28 through Day 196 or used any additional antipseudomonal antibiotics from Day 28 through Day 196.
Arm/Group | AZLI - Sensitivity Analysis Set
Number analyzed (Participants) | 98
percentage of participants | 46.9 [37.1 to 56.8]

ADVERSE EVENTS:
Time Frame: Baseline to Day 28 plus 30 days
Groups:
- AZLI: Treatment-emergent adverse events and treatment-emergent serious adverse events were collected from Baseline through Day 28 plus 30 days.
  Participants received one 28-day course of AZLI, then were followed for a 24-week period (through Day 196). AZLI 75 mg was administered 3 times daily via the investigational eFlow® nebulizer.
Arm/Group | AZLI
Serious Adverse Events (participants affected / at risk) | 8/105
Other Adverse Events (participants affected / at risk) | 66/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI (N=105)
Hepatitus acute (Hepatobiliary disorders) | 1
Infectious mononucleosis (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 1
Pseudomonas test positive (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI (N=105)
Diarrhoea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Pyrexia (General disorders) | 15
Rhinitis (Infections and infestations) | 8
Pseudomonas test positive (Investigations) | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 42
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years